CLINICAL TRIAL: NCT05974852
Title: Effect of Ocrelizumab on Choroid Plexus Changes in Patients With Primary-progressive Multiple Sclerosis Participating in the ORATORIO: a Post-hoc Analysis of a Double-blind, Randomized, Phase 3, Placebo-controlled Study
Brief Title: Effect of Ocrelizumab on Choroid Plexus Changes in Patients With PPMS
Acronym: ORATORIO-CP
Status: Active, not recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Principal Investigator, State University of New York at Buffalo
Other Study IDs: 00007537
Record Dates: First submitted 2023-07-12; First posted 2023-08-03 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Primary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Ocrelizumab — Non-interventional

SUMMARY:
The goal of this non-interventional, observational study is to learn if cortical plexus enhancement in patients with primary progressive multiple sclerosis occurs in response to the autoimmune inflammatory process.

DETAILED DESCRIPTION:
To study the effect of ocrelizumab on choroid plexus changes in patients with primary-progressive multiple sclerosis participating in the ORATORIO: a post-hoc analysis of a double-blind, randomized, phase 3, placebo-controlled study

ELIGIBILITY:
Inclusion Criteria:

* Patient participating in the ORATORIO study
* MRI scans available at baseline
* Presence of T2-weighted image (WI) (FLAIR, T2/PD), and 3D T1-WI at baseline

Exclusion Criteria:

- None

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with primary progressive multiple sclerosis
Sampling Method: Non-Probability Sample
Enrollment: 732 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
T2 lesion volume | 5 years
  T2 lesion volume as measured using MRI.

SECONDARY OUTCOMES:
Changes in choroid plexus | 5 years
  Changes in choroid plexus as measured using MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Buffalo Neuroimaging Analysis Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No